CLINICAL TRIAL: NCT03854799
Title: Phase II Study Of Preoperative Chemoradiotherapy Plus Avelumab In Patients With Locally Advanced Rectal Cancer
Brief Title: Immunotherapy In Locally Advanced Rectal Cancer
Acronym: AVANA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-003582-10
Record Dates: First submitted 2019-02-12; First posted 2019-02-26 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Colon Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — avelumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHEMORADIOTHERAPY PLUS AVELUMAB (Experimental): CHEMORADIOTHERAPY PLUS AVELUMAB:
  CAPECITABINE 825 mg/sqm/bid p.o. 5 days/week EXTERNAL-BEAM IRRADIATION 50.4 GY in 28 fractions over 5.5 weeks AVELUMAB 10 mg/Kg ev over 1 hour every 2 weeks at days 1, 14, 28, 42, 56, 70
  Interventions: Drug: Avelumab; Drug: Capecitabine; Radiation: EXTERNAL---BEAM IRRADIATION 50.4 GY

INTERVENTIONS:
Drug: Avelumab — Eligible patients will receive:
  CHEMORADIOTHERAPY PLUS AVELUMAB:
  * CAPECITABINE 825 mg/sqm/bid p.o. 5 days/week
  * EXTERNAL-BEAM IRRADIATION 50.4 GY in 28 fractions over 5.5 weeks
  * AVELUMAB 10 mg/Kg ev over 1 hour every 2 weeks at days 1, 14, 28, 42, 56, 70
  Surgery with TME must be performed at week 8-10 after the end of CTRT. The final choice of surgical procedure (ie, abdominoperineal surgery or anterior resection) is at the surgeon's discretion.
Drug: Capecitabine — Eligible patients will receive:
  CHEMORADIOTHERAPY PLUS AVELUMAB:
  * CAPECITABINE 825 mg/sqm/bid p.o. 5 days/week
  * EXTERNAL-BEAM IRRADIATION 50.4 GY in 28 fractions over 5.5 weeks
  * AVELUMAB 10 mg/Kg ev over 1 hour every 2 weeks at days 1, 14, 28, 42, 56, 70
  Surgery with TME must be performed at week 8-10 after the end of CTRT. The final choice of surgical procedure (ie, abdominoperineal surgery or anterior resection) is at the surgeon's discretion.
Radiation: EXTERNAL---BEAM IRRADIATION 50.4 GY — Surgery with TME must be performed at week 8-10 after the end of CTRT. The final choice of surgical procedure (ie, abdominoperineal surgery or anterior resection) is at the surgeon's discretion.

SUMMARY:
Preoperative CTRT is considered the standard of care in the management of LARC. Preoperative CTRT approach results in significant tumor downstaging and local control with a complete pathological response rate of about 15% even if additional therapeutic strategies should be explored to improve outcomes, expecially for T4 cancers.

Immunotherapy with PD-1/PD-L1 immunocheckpoint blockade (ICB), turned out a breakthrough in cancer treatment among different tumor types, including CRC. An ICB strategy could lead up to a 40% of response in metastatic CRC with deficient mismatch repair (MMR) status. Unfortunately, the activity of ICBs in MMR proficient mCRC is extremely low but it might be improved using immunomodulatory strategies as demonstrated by Bendell et al.

In this context, the role of RT in revert the tolerance to a low neoantigen-burden (such as in MMR proficient CRCs) by the induction of antigen release from the tumour and activation of dendritic cells leading to a CD8+ T lymphocyte-mediated anticancer immune response has been widely elucidated. Moreover, antineoplastic agents can be exploited to target other crucial cellular effectors of immunosuppressive tumor microenvironment (i.e. regulatory T cells and myeloid-derived suppressor cells).

In line with these evidences, Hecht et al. have recently reported that in rectal cancer patients, neoadjuvant CTRT increases PD-L1 expression in tumor cells, strongly suggesting a neoadjuvant combinatory strategy with RT and PD-1/PD-L1 pathway blockade. The integration of immunotherapy in the neoadjuvant setting (instead of adjuvant one) for the management of LARC is also supported by preclinical findings showing that in metastatic breast cancer mice models, neoadjuvant immunotherapy is superior in inducing long-term survivors, compared with adjuvant strategy with a greater magnitude of tumor-specific T cell expansion in neoadjuvant treated mice and a better anti-tumor T cell-mediated immune response.

On the basis of such considerations, there is a strong biological and clinical rationale for testing the addition of avelumab, an anti-PD-L1 moab, to capecitabine-based CTRT in patients with technically resectable, LARC. The aim of this strategy is to lead to significant improvements of pCR and, ultimately, patients' survival.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to study procedures.
* Histologically proven diagnosis of rectal adenocarcinoma
* Locally advanced, resectable disease defined by the presence of at least one of the following features:

  * cN+ (with the definition of a clinically positive lymph node being any node ≥ 1 cm)
  * cT4
  * high risk cT3 (according to magnetic resonance imaging [MRI] criteria): tumour extending to within 1 mm of or beyond the mesorectal fascia (ie, circumferential radial margin threatened or involved); lower third (≤ 6 cm from the anal verge); tumour extending 5 mm or more into perirectal fat
* Distal tumor margin at < 12 cm from the anal verge
* No evidence of metastatic disease by computed tomography (CT) scan of the chest and abdomen and total body FDG-PET/CT scan
* Tumor must be amenable to curative resection (curative resection can include pelvic exenteration)
* No history of invasive rectal malignancy, regardless of disease-free interval
* No other rectal cancers (i.e., sarcoma, lymphoma, carcinoid, squamous cell carcinoma, or cloacogenic carcinoma) or synchronous colon cancer
* No clear indication of involvement of the pelvic side walls by imaging
* Age ≥ 18 years
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1
* Life expectancy of at least 5 years (excluding diagnosis of cancer)
* Hematopoietic: absolute neutrophil count ≥ 1,500/mm3; platelet count ≥ 100,000/mm3; haemoglobin level ≥ 9 g/dL
* Hepatic: total bilirubin ≤ 1.5 times upper limit of normal (ULN); alkaline phosphatase ≤ 2 times ULN; AST and ALT ≤ 2.5 times ULN [Note: *If AST>ULN, serologic testing for Hepatitis B and C must be negative]
* Renal: creatinine clearance ¬≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method); no renal disease that would preclude study treatment or follow-up
* Available tumor samples at baseline (archival biopsy) and after chemoradiotheraphy + avelumab
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception as outlined in Section 5.5 - Contraception, starting with the first dose of study therapy through 180 days after the last dose of treatment Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Women of childbearing potential must have a negative blood or urine pregnancy test at the baseline visit
* Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.5 - Contraception, for the course of the study starting with the first dose of study therapy through 180 days after the last dose of treatment Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject
* Will and ability to comply with the protocol.

Exclusion Criteria:

* Previous therapy with any antibody or drug targeting T cell coregulatory proteins, or immunosuppressive agents
* Previous pelvic RT
* Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible
* Any of the following in the 6 months prior to treatment start: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, congestive heart failure (≥ New York Heart Association Classification Class II), cerebrovascular accident/strock, transient ischemic attack, serious cardiac arhythmia requiring medication or symptomatic pulmonary embolism
* Uncontrolled coagulopathy
* Active infection requiring systemic therapy
* Current use of immunosuppressive medication, EXCEPT for the following: a. Intranasal, inhaled, topical steroids, or local steroids injection (e.g. intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Prior organ transplantation including allogenic stem-cell transplantation
* Active tubercolosis
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive)
* Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3)
* Pregnant female patients, breastfeeding female patients, and male patients able to father children and female patients of childbearing potential who are unwilling or unable to use 2 highly effective methods of contraception as outlined in the protocol for the duration of the study
* Lack of upper gastrointestinal tract integrity or malabsorption syndrome; immune colitis; active inflammatory bowel disease (i.e., patients requiring current medical interventions or who are symptomatic)
* Patients with prior malignancies (with the exception of rectal cancer), including invasive colon cancer, are eligible provided they have been disease-free for ≥ 5 years and are deemed by their physician to be at low risk for recurrence
* Other malignancy within the past 5 years with the exception of effectively treated squamous cell or basal cell skin cancer, melanoma in situ, carcinoma in situ of the cervix, or carcinoma in situ of the colon or rectum
* Other severe acute or chronic medical conditions including immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies.
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study and until 180 days after the last trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The primary objective of this trial is to evaluate the rate of complete pathologic response (pCR) | 24 months
  pCR rate is defined as the percentage of patients, relative to the total of enrolled subjects,achieving complete histological regression with no available tumor cells yT0N0

SECONDARY OUTCOMES:
R0 resection rate | 24 months
  is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing R0 resection of primary tumour
Tumor downstaging | 24 months
  is defined as reduction of at least one level in T or N staging between the baseline MRI and histopathological staging, without evidence of upstaging or disease progression.
Local recurrence | 24 months
  is defined as an intrapelvic recurrence following a primary rectal cancer resection, with or without distal metastasis.
Sphincter preservation rate | 24 months
  is defined as the percentage of patients undergoing sphincter-sparing surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No